CLINICAL TRIAL: NCT05653011
Title: Predictors of Response After Induction Therapy With TNF-alpha Inhibitor in Inflammatory Bowel Disease, Comparison to Normal
Brief Title: Predictors of Prognosis in IBD Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nayoung Kim, professor, Seoul National University Bundang Hospital
Other Study IDs: B-1305-201-001
Record Dates: First submitted 2022-10-25; First posted 2022-12-15 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Disease
Keywords: inflammatory bowel disease; ulcerative colitis; crohn's disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — endoscopically biopsied sample blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Control group: Patients who are not diagnosed with inflammatory bowel disease and have colitis.
  Interventions: Other: Endoscopic biopsy
- TNF-alpha Inhibitor-naive IBD group: Patients who are diagnosed with inflammatory bowel disease but do not have a history of TNF-a inhibitor treatment.
  Interventions: Other: Endoscopic biopsy
- TNF-alpha Inhibitor-treated IBD group: Patients who are diagnosed with inflammatory bowel disease and have a history of TNF-a inhibitor treatment.
  Interventions: Other: Endoscopic biopsy

INTERVENTIONS:
Other: Endoscopic biopsy — When patients have colonoscopy or sigmoidoscopy for evaluation of their disease course, biopsied samples are collected.
  In the IBD group, samples are obtained at endoscopically active and/or inactive lesions. In the control group, samples are obtained at endoscopically normal lesions.

SUMMARY:
A study of clinical characteristics and potential prognostic factors in inflammatory bowel disease

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is a chronic and relapsing inflammatory disease composed of two types: Crohn's disease (CD) and ulcerative colitis (UC). It is difficult to cure the IBD completely and patients with clinical or endoscopic remission can worsen again. Therefore, predicting the prognosis of patients with IBD is still challenging.

Endoscopic biopsied samples and blood samples from IBD patients and non-IBD controls have been collected and the expression levels of multiple markers which are associated with disease activity and severity will be assessed. The correlation between expression levels of multiple markers and prognosis will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* control group: Patients who do not have colitis, cancer, and advanced polyp (the number of polyps ≥ 3, the size of polyps ≥ 1cm, high-grade adenoma, villous adenoma)
* TNF-α inhibitor-naive IBD group: IBD patients who do not have a history of TNF-α inhibitor treatment
* TNF-α inhibitor-treated IBD group: IBD patients who are treated with TNF-α inhibitor

Exclusion Criteria:

* Age under 18 years
* Patients who were treated with antibiotics or probiotics within the last 3 months

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who visited Seoul National University Bundang Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-03-11 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The expression level of multiple markers associated with IBD activity or prognosis | baseline (at the time of enrollment)
  The expression level of multiple markers was evaluated through RT-qPCR using endoscopically biopsied samples or blood samples. Markers include TGF-b, SLUG, SNAIL, E-cadherin, vimentin, OLFM4, LGR5, a-SMA, FSP1, IL-17A, IL-23, TGF-b, IL-6, IFN-r, IL-1b, FOXP3, PD-1, CD68, PAD4, COL3A1, TIMP3, LOX, ACTA2, ITGB6, CAV-1 etc.

SECONDARY OUTCOMES:
The change of expression level of multiple markers associated with IBD activity or prognosis | Every 2 years. The examination will be suspended when treatment was ended.
  The change of expression level of multiple markers was evaluated through RT-qPCR using endoscopically biopsied samples or blood samples. Markers include TGF-b, SLUG, SNAIL, E-cadherin, vimentin, OLFM4, LGR5, a-SMA, FSP1, IL-17A, IL-23, TGF-b, IL-6, IFN-r, IL-1b, FOXP3, PD-1, CD68, PAD4, COL3A1, TIMP3, LOX, ACTA2, ITGB6, CAV-1 etc. (compared to results 2 year ago)

CONTACTS AND LOCATIONS:
Overall Officials: Nayoung Kim, M.D., Ph.D, Study Chair — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jun YK, Kim N, Yoon H, Park JH, Kim HK, Choi Y, Lee JA, Shin CM, Park YS, Lee DH. Molecular Activity of Inflammation and Epithelial-Mesenchymal Transition in the Microenvironment of Ulcerative Colitis. Gut Liver. 2024 Nov 15;18(6):1037-1047. doi: 10.5009/gnl230283. Epub 2024 Feb 22. PMID 38384179